CLINICAL TRIAL: NCT00536640
Title: Inoperable Non-Squamous NSCLC Stage III/IV: A Randomised Phase II Study With Bevacizumab Plus Erlotinib Or Gemcitabin/Cisplatin Plus Bevacizumab
Brief Title: Inoperable Non-Squamous NSCLC Stage III/IV: A Randomised Phase II Study With Bevacizumab Plus Erlotinib Or Gemcitabine/Cisplatin Plus Bevacizumab
Acronym: INNOVATIONS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aktion Bronchialkarzinom e.V. (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABC-2006-NSCLC-01; 2006-004865-32 (EudraCT Number)
Record Dates: First submitted 2007-09-27; First posted 2007-09-28 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Non Small Cell Lung Carcinoma (NSCLC Stage III an IV)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Bevacizumab; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Erlotinib, Bevacizumab) (Experimental)
  Interventions: Drug: Erlotinib; Drug: Bevacizumab
- Arm B (Gemcitabine, Cisplatin, Bevacizumab) (Active Comparator)
  Interventions: Drug: Bevacizumab; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Erlotinib — 150 mg per os, given daily until tumor progression
  Arms: Arm A (Erlotinib, Bevacizumab)
Drug: Bevacizumab — 15mg/kg i.v. on day 1 (three-week cycle) until tumor progression
Drug: Gemcitabine — 1250 mg/2 i.v. on day 1 and day 8 (three-week cycle) until tumor progression for a maximum of 6 cycles
  Arms: Arm B (Gemcitabine, Cisplatin, Bevacizumab)
Drug: Cisplatin — 80 mg/m2 i.v. on day 1 (three-week cycle) until tumor progression for a maximum of 6 cycles. (The administration of 40 mg/2 Cisplatin on day 1 and day 8 is also possible)
  Arms: Arm B (Gemcitabine, Cisplatin, Bevacizumab)

SUMMARY:
This study wants to determine the activity of a non chemotherapy first line biological treatment with Erlotinib/Bevacizumab or Gemcitabine-Cisplatin/Bevacizumab in patients with the diagnosis of non-squamous advanced Non Small Lung Cancer.

DETAILED DESCRIPTION:
Prospective, randomized multi-center, open label phase II study to determine the activity of a non-chemotherapy first line biological treatment with Erlotinib/Bevacizumab or Gemcitabine-Cisplatin/Bevacizumab in patients with the diagnosis of non-squamous advanced Non-Small-Lung-Cancer.

* Duration of treatment/patient: up to 1,5 years
* Follow Up: ≈ 6 month
* Planned number of patients: 220 treated patients (110 patients/arm)

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmed Non-Small Cell Lung Cancer that can not be treated within a defined radiological field
* Tumor stage IIIB (pleural effusion or pericardial effusion included) or IV
* The following histological tumor types are eligible:

  * Adenocarcinoma (including adenocarcinomas with bronchioloalveolar differentiation)
  * Large Cell Carcinoma (including large cell carcinomas with neuroendocrine differentiation)
  * Mixed Cell Carcinoma without small cell fraction and without predominant squamous cell fraction (< 50%)
  * undifferentiated non-small-cell-carcinoma
* No previous chemotherapy within the last five years
* At least 4 weeks since last major surgery
* Age ≥ 18 years
* ECOG <= 2
* Adequate hematological laboratory parameters

  * Hemoglobin ≥ 10 g/dl
  * WBC ≥ 3.000/µl
  * Platelets ≥ 100.000/µl
* Adequate hepatic laboratory parameters

  * Bilirubin <= 2,0 mg/dl
  * AST(GOT) <= 2,5 x ULN in patients without liver metastases
  * AST(GOT) <= 5 x UNL in patients with liver metastases
  * ALT(GPT) <= 2,5 x ULN in patients without liver metastases
  * ALT(GPT) <= 5 x UNL in patients with liver metastases
* Adequate renal laboratory parameters

  * Creatinine <= 1,5 mg/dl
  * Creatinine Clearance > 60 ml/min
* Adequate plasmatic blood coagulation - INR <= 1,5 and PTT <= 1,5 x ULN
* Normal cardiac function defined by LVEF > 49% (echocardiography)
* Electrocardiogram without significant signs of cardiac arrhythmias
* Provision of informed consent according to local regulatory requirements prior to any protocol specific treatment
* Measurable lesion according to RECIST-Criteria's
* Negative pregnancy test for women of childbearing potential unless they are postmenopausal at baseline. (Postmenopausal women must have been amenorrheic at least for 12 months to be considered of non childbearing potential)
* Women of child bearing potential to must be willing to use an acceptable method to avoid pregnancy at least one month before study start. Examples: oral contraceptives (sole application of oral contraceptives is not sufficient), diaphragm pessary, intrauterine device (spiral), condom plus diaphragm pessary plus spermicide

Exclusion Criteria:

* Histologic confirmed squamous cell carcinoma
* Pregnancy or lactation period
* Tumor extension treatable with radiotherapy
* Current clinical signs or symptoms of brain and/or leptomeningeal metastases confirmed by CT or MRI brain scan
* Evidence of tumor invading or abutting major blood vessels
* Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of a CIS of the cervix or non-melanomatous skin cancer. Patients curatively treated and free of disease for at least 5 years will be discussed with the Principal Investigator (LKP) before inclusion
* Any previous chemotherapy within the last five years
* Any radiotherapy with exception of the following situations:

  * concomitant small field radiotherapy in the case of solitary bone metastases or other solitary metastases
  * in case of large field radiotherapy or multi-radiation fields due to multiple bone metastases or other metastases. The application of study medication then must be delayed at least for 24 h (after last radiotherapy)
  * in case of radiotherapy of the primary tumor trial therapy can be employed if radiotherapy has ended at least 6 weeks ago and new tumor progression is clearly documented
* Treatment with an investigational new drug, currently or within the last 28 days, and/or participation in another clinical trial, currently or during the last 12 weeks, and/or previous participation in this study
* A history or presence of any CNS disorder or psychiatric disability judged by the Investigator to be clinically significant and/or interfering with compliance of oral drug intake
* Patients with any clinically significant disease that in the opinion of the investigator is likely to put the patient at risk or to interfere with the evaluation of the patient's safety and of the study outcome. This includes, but is not limited to:

  * Any known significant ophthalmologic abnormalities of the surface of the eye (the use of contact lenses is not recommended)
  * Immediate need for therapeutic intervention (e.g.: upper inflow congestion or poststenotic pneumonia)
  * Clinically significant cardiac disease (e.g. right-sided heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 6 months
  * pleural effusion or pericardial effusion with the need for intervention
* Uncontrolled hypertension
* Non healing wound, ulcer or bone fracture
* Fresh thrombosis under therapy with anticoagulants
* Hemorrhagic diathesis, Hemophilia A, Hemophilia B
* Implantation of a central vein catheter (Prot-Catheter) within 24 h prior to application of study medication
* Present hemoptysis of any CTC grade or history of hemoptysis of any CTC grade within 3 month prior to study start
* Peritoneal carcinomatosis
* History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 month prior to study start
* Interstitial pneumonia or extensive or symptomatic interstitial fibrosis of the lung
* Pleural effusion or ascites, which cause respiratory compromise
* Any other active or uncontrolled infection
* Organ allograft
* History of a mental disease or condition such as to interfere with the patient's ability to understand the requirements of the study and the intake of study medication according to study protocol
* Inability to swallow pills
* Current or recent (within 10 days of first dose of study medication) use of coumadin/warfarin or marcumar/phenprocoumon for therapeutic purposes Prophylactic use of low molecular weight heparins is allowed
* Current or recent (within 10 days of first dose of study medication) use of ASS - Dosage > 325 mg/day
* Current or recent (within 10 days of first dose of study medication) use of Plavix/Clopidogrel
* Alcohol and drug abuse
* Known hypersensitivity to any of the study drugs
* Presence of a tracheobronchial fistula or fistulization in other organ systems like gastrointestinal fistulas or fistulization of urogenital tract

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2007-11; Primary Completion 2011-08 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
The main efficacy parameter is the progression free survival. | Recruitment 1 year, Follow up 2 years

SECONDARY OUTCOMES:
Overall survival | Recruitment 1 year, Follow up 2 years
Quality of life | Screening, prior to next treatment cycle, treatment day 126, end of therapy
Response rate | Screening, prior to treatment cycle 3, prior to treatment clycle 5, treatment day 126, every 6 weeks after treatment day 126, end of therapy
Molecular investigations | Screening, prior to treatment cycle 3

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Martin Wolf, MD, Principal Investigator — Aktion Bronchialkarzinom e.V.
Locations (37):
- Germany (37):
  - Klinikum Bayreuth GmbH, Bayreuth
  - Charite´ Mitte, Berlin
  - Gemeinschaftskrankenhaus Havelhöhe, Berlin
  - Helios Klinikum Emil v. Behring, Berlin
  - Augusta-Krankenanstalten, Bochum
  - Johanniter-Krankenhaus Bonn, Bonn
  - Forschungszentrum Borstel, Borstel
  - Malteser Krankenhaus St. Hildegardis, Cologne
  - St. Johannes Hospital, Duisburg
  - Städtisches Krankenhaus Frankfurt-Höchst, Frankfurt
  - Klinikum Frankfurt (Oder)GmbH, Frankfurt (Oder)
  - Krankenhaus Nordwest, Frankfurt am Main
  - Medizinisches Versorgungszentrum Osthessen, Fulda
  - Georg-August-Universität Göttingen, Göttingen
  - Universitätsklinikum Greifswald, Greifswald
  - Krankenhaus Großhansdorf, Großhansdorf
  - Diakoniekrankenhaus Halle/S., Halle
  - Asklepios Klinik Harburg, Hamburg
  - Thoraxklinik Universitätsklinikum Heidelberg, Heidelberg
  - Lungenklinik Hemer, Hemer
  - Fachklinik für Lungenerkrankungen Immenhausen, Immenhausen
  - St. Vincentius-Kliniken Karlsruhe, Karlsruhe
  - Klinikum Kassel GmbH, Kassel
  - Katholisches Klinikum Haus Marienhof, Koblenz
  - Onkologische Schwerpunktpraxis Dr. Lothar Müller, Leer
  - Klinikum Lippe-Lemgo, Lemgo
  - Klinik Löwenstein, Löwenstein
  - Klinikum Ludwigshafen, Ludwigshafen
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - St. Hildegardis Krankenhaus, Mainz
  - Universitätsklinikum Marburg, Marburg
  - Johannes Wesling Klinikum Minden, Minden
  - Krankenhaus Barmherzige Brüder, Regensburg
  - Hanse-Klinikum Stralsund, Stralsund
  - Onkologische Gemeinschaftspraxis Dr. Nusch, Velbert
  - Fachkliniken Wangen, Wangen
  - Helios Klinikum Wuppertal, Wuppertal

REFERENCES:
- [Derived] Thomas M, Fischer J, Andreas S, Kortsik C, Grah C, Serke M, von Eiff M, Witt C, Kollmeier J, Muller E, Schenk M, Schroder M, Villalobos M, Reinmuth N, Penzel R, Schnabel P, Acker T, Reuss A, Wolf M; ABC-Lung Cancer Group. Erlotinib and bevacizumab versus cisplatin, gemcitabine and bevacizumab in unselected nonsquamous nonsmall cell lung cancer. Eur Respir J. 2015 Jul;46(1):219-29. doi: 10.1183/09031936.00229014. Epub 2015 Mar 18. PMID 25792638